CLINICAL TRIAL: NCT04342858
Title: A Prospective Randomized Controlled Trial for Prevention of Enamel White Spot Lesions During Fixed Orthodontic Treatment
Brief Title: Prospective Randomized Controlled Trial for Prevention of Demineralization During Fixed Orthodontic Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Version no.3; 27th Nov'17
Record Dates: First submitted 2020-04-02; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Demineralization, Tooth; Caries,Dental; White Spot Lesion
Keywords: orthodontics; demineralizatiion; fluoride; Diagnodent
MeSH Terms: conditions — Tooth Demineralization; Dental Caries | interventions — tricalcium phosphate; Health Education, Dental

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with three parallel groups. In the proposed study, individual participants, and not parts of the mouth, will serve as the unit of randomization. This approach unlike a split-mouth design will eliminate the problems of cross-contamination.
Who Masked: Participant, Outcomes Assessor
Masking Description: A dental assistant will allocate the participants in the study to their respective groups. The examiner will not be informed about the study participant's group allocation information. The orthodontist performing the fixed orthodontic treatment will not know about the study participant's group allocation information as the topical fluoride varnish application in this study will be performed by another operator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (Other): Control will receive standard oral hygiene instructions (OHI every three months)
  Interventions: Other: Oral health education
- Standard of care + Fluoride varnish (Active Comparator): Intervention 1 will receive standard OHI and application of topical fluoride varnish containing 5% NaF (Duraphat varnish®, Colgate-Palmolive (UK) Ltd., Guildford, Surrey, UK) every three months
  Interventions: Drug: Fluoride Varnish
- Standard of care + Fluoride varnish with Tricalcium phosphate (Experimental): Intervention 2 will receive standard OHI and application of topical fluoride varnish containing 5% NaF + TCP (Clinpro white varnishTM, 3M ESPE, St Paul, MN, USA) every three months
  Interventions: Drug: Fluoride Varnish with tricalcium phosphate

INTERVENTIONS:
Drug: Fluoride Varnish — Duraphat varnish®, Colgate-Palmolive (UK) Ltd., Guildford, Surrey, UK
  Other Names: 5% Sodium fluoride varnish
  Arms: Standard of care + Fluoride varnish
Drug: Fluoride Varnish with tricalcium phosphate — Clinpro white varnishTM, 3M ESPE, St Paul, MN, USA
  Other Names: 5% Sodium fluoride varnish containing tri-calcium phosphate
  Arms: Standard of care + Fluoride varnish with Tricalcium phosphate
Other: Oral health education — Standard oral hygiene instructions every 3 months
  Other Names: Oral hygiene instructions
  Arms: Standard of care

SUMMARY:
Treatment with fixed orthodontic appliances is often associated with pain, which poses great challenges in the efficient brushing of the teeth thus making the teeth more vulnerable to plaque formation. Treatment duration with fixed orthodontic appliances usually extends to 18 months or even longer in some cases. This prolonged vulnerability to plaque formation frequently leads to demineralization of teeth. There is also an increase in the number of plaque retentive sites due to the fixed appliances, leading to a rapid change in the bacterial composition of the dental plaque, particularly in the number of acidogenic bacteria. The resulting enamel decalcification is also known as white spot lesions (WSLs), which is an early sign of demineralization of enamel. Enamel WSLs (EWSLs) can be observed even as early as four weeks from the start of fixed orthodontic treatment. The occurrence of EWSLs adjacent to the orthodontic brackets ranges from 15 to 85%.

The incidence of EWSLs development is higher in orthodontic patients as compared to the development of similar lesions in non-orthodontic patients. These EWSLs are not aesthetically pleasing and is certainly unacceptable when it develops during fixed orthodontic treatment that is usually performed in patients who often seek such treatment to improve their aesthetics. Additionally, even if the outcome of fixed orthodontic treatment is superior from well-aligned teeth, aesthetics can be greatly compromised with EWSLs. Therefore, the prevention of such lesions is an important concern for orthodontists.

Though professionally applied topical fluoride varnish helps in remineralization of EWSLs, an adequate supply of calcium and phosphate ions is essential for remineralization. Therefore, EWSLs on maxillary teeth could be prevented and remineralized by the use of advanced novel topical fluoride varnish with added calcium and phosphate-based delivery system.

DETAILED DESCRIPTION:
Fluoride is proven caries preventive and therapeutic agent. It helps in the remineralization of early enamel caries lesions and subsequently increases its resistance to dissolution by acids produced by cariogenic microflora. Topical fluoride varnish was introduced in the 1960s. The Food and Drug Administration (FDA) in the USA approved the use of fluoride varnishes for dentistry in 1994 and presently fluoride varnish is the most commonly used professionally applied topical fluoride agent. The most popular topical fluoride varnish is Duraphat®, which contains 5% NaF varnish (2.2% Fluoride). The greatest advantage of topical fluoride varnish is its ability to adhere to tooth tissues for a longer period of time that enables improved fluoride uptake. It allows the continuous release of fluoride ions into enamel, dentine, plaque, and saliva. Additionally, the application of topical fluoride varnish is a simple procedure and does not require great patient co-operation. Topical fluoride varnish application has been reported to exhibit substantial caries inhibiting effect in both permanent and primary teeth.

Among the various forms of fluoride products, such as gels, varnishes, foams, mouth- rinses, and toothpastes, varnishes do not rely on patient compliance and cooperation. The major advantage of varnishes is high retention followed by gradual release of fluoride over an extended time period, which leads to low concentrations in the liquid plaque-enamel interface. The use of fluoride diminishes demineralization and promotes remineralization, thereby balancing the process of caries formation. A recent Cochrane review has revealed moderate evidence for the prevention of EWSLs during fixed orthodontic treatment by fluoride varnish application every six weeks at the time of orthodontic review, but this finding is based on a single study. Therefore, the quality of the evidence found is moderate and the review recommendations state that additional well- conducted research is required in this area.

Caries preventive and inhibiting effect of topical fluoride therapy depends on an adequate supply of calcium and phosphate ions. Though calcium and phosphate ions are supplied naturally by saliva, the concentration of such ions is low (even lower in patients suffering from reduced salivary flow). Low concentration of salivary calcium and phosphate ions leads to a mineral deposition only at the surface of the enamel as a result of a low ion concentration gradient. The deposition of minerals at the surface of enamel alone may not improve the structural properties of the deeper part of the early-stage or incipient caries lesions. This has led to the introduction of calcium phosphate-based delivery systems containing high concentrations of calcium phosphate such as tri-calcium phosphate (TCP).

Tri-calcium phosphate (TCP) is a product resulting from ball milling beta-tri-calcium phosphate with sodium lauryl sulphate. ClinproTM white varnish (3M ESPE, St Paul, MN, USA), which contains TCP and NaF, is a commercially available topical fluoride varnish, which claims that the protective fumaric acid barrier facilitates co-existence of calcium and fluoride ions, however, during storage, the unwanted reaction between the ions is prevented. The protective barrier breaks upon contact with saliva, releasing the ions for effective remineralization of the tooth. At present there is no clinical study to prove the superior EWSLs-preventive effect of this newer NaF varnish with TCP when compared to conventional topical NaF varnish in patients undergoing fixed orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects about to undergo multi-bracketed fixed orthodontic treatment will be invited to participate in this study.

Exclusion Criteria:

1. History of fixed orthodontic treatment
2. Presence of any developmental defects of enamel (DDE) on labial surfaces of teeth
3. Presence of any dental anomalies or direct/indirect labial restorations on teeth
4. History of long-term antibiotic usage
5. Presence of untreated cavitated lesions
6. Plaque level greater than 25%
7. Patients requiring complicated orthognathic surgeries

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Enamel White Spot Lesions index surface scores: Clinical evaluation (Subjective criteria) | 24 months
  Changes in EWSLs surface scores (using Gorelick's index, 1982) among three study groups (evaluated clinically).
  The Gorelick's index is graded as: 0 (no lesion), 1(moderate lesion), 2 (severe lesion) and 3 (cavitation) with lower score representing good outcome and higher score representing poor outcome.
Change in Enamel White Spot Lesions index surface scores: Photographic evaluation (Subjective criteria) | 24 months
  Changes in EWSLs surface scores (using Gorelick's index, 1982) among three study groups (evaluated photographically).
  The Gorelick's index is graded as: 0 (no lesion), 1(moderate lesion), 2 (severe lesion) and 3 (cavitation) with lower score representing good outcome and higher score representing poor outcome
Change in Laser fluoroscence values (Objective criteria) | 24 months
  Changes in mean DIAGNOdent scores among three study groups. The DIAGNOdent values (or laser fluorescence values) are visible on the device as digital readings from 0 to 99 with higher readings representing poor outcomes and lower readings representing good outcomes.

SECONDARY OUTCOMES:
Enamel White Spot Lesions index surface scores: Clinical evaluation (Subjective criteria) | 6 months
  EWSLs surface scores (using Gorelick's index, 1982) among three study groups (evaluated clinically)
Enamel White Spot Lesions index surface scores: Clinical evaluation (Subjective criteria) | 12 months
  EWSLs surface scores (using Gorelick's index, 1982) among three study groups (evaluated clinically)
Enamel White Spot Lesions index surface scores: Clinical evaluation (Subjective criteria) | 18 months
  EWSLs surface scores (using Gorelick's index, 1982) among three study groups (evaluated clinically)
Enamel White Spot Lesions index surface scores: Photographic evaluation (Subjective criteria) | 6 months
  EWSLs surface scores (using Gorelick's index, 1982) among three study groups (evaluated photographically)
Enamel White Spot Lesions index surface scores: Photographic evaluation (Subjective criteria) | 12 months
  EWSLs surface scores (using Gorelick's index, 1982) among three study groups (evaluated photographically)
Enamel White Spot Lesions index surface scores: Photographic evaluation (Subjective criteria) | 18 months
  EWSLs surface scores (using Gorelick's index, 1982) among three study groups (evaluated photographically)
Laser fluoroscence evaluation (Objective criteria) | 6 months
  Mean DIAGNOdent scores among three study groups
Laser fluoroscence evaluation (Objective criteria) | 12 months
  Mean DIAGNOdent scores among three study groups
Laser fluoroscence evaluation (Objective criteria) | 18 months
  Mean DIAGNOdent scores among three study groups

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia KY Yiu, MDS, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Data Management Plan (DMP) has been submitted to the university repository and final data will be deposited to the university.